CLINICAL TRIAL: NCT03576664
Title: Effects of Sleep Deprivation and Adrenergic Inhibition on Glymphatic Flow in Humans
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Gitte Moos Knudsen (Other)
Collaborators: University of Copenhagen (Other); Danish Center for Sleep Medicine (Other)
Responsible Party: Sponsor-Investigator, Gitte Moos Knudsen, Center director of Center for Integrated Molecular Brain Imaging, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: sleepgf; H-16045933 (Other: Ethical Committee)
Record Dates: First submitted 2018-03-08; First posted 2018-07-03 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Sleep Deprivation; Sleep Wake Disorders; Sleep
Keywords: carvedilol; adrenergic antagonists; glymphatic system; volunteers; Molecular Mechanisms of Pharmacological
MeSH Terms: conditions — Sleep Deprivation; Sleep Wake Disorders | interventions — Carvedilol

STUDY DESIGN:
Intervention Model Description: Randomized, cross-over, placebo-controlled study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carvedilol first (Experimental): Carvedilol (25 mg) followed by Placebo oral capsule is administered in a crossover manner.
  Interventions: Drug: Carvedilol 25mg; Drug: Placebo oral capsule
- Placebo first (Experimental): Placebo oral capsule followed by Carvedilol (25 mg) is administered in a crossover manner.
  Interventions: Drug: Carvedilol 25mg; Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Carvedilol 25mg — Cross-over, randomized, placebo-controlled study.
  Other Names: Coreg
Drug: Placebo oral capsule — Cross-over, randomized, placebo-controlled study.

SUMMARY:
The project is aimed at identifying how the adrenergic antagonist 'carvedilol' modulates the effects of sleep deprivation in healthy volunteers. The study is a double-blind, randomized, placebo-controlled, cross-over study. Investigators will include 20 healthy volunteers who will undergo three functional magnetic resonance (fMRI) imaging sessions, one at baseline, and two after sleep deprivation (one night without sleep). The two sleep-deprivation scans are performed in a randomized order where subjects receive placebo or carvedilol, in a within-subject, cross-over study design.

The following domains will be described: 1) fMRI imaging of cerebrospinal fluid (CSF) pulsations (glymphatic flow) in the human brain, performed by a combination of fMRI protocols that includes structural (T1, T2, diffusion weighted) and functional (multiband/fast imaging, spectroscopy) imaging. 2) fMRI imaging during wakefulness and sleep are determined by simultaneous electroencephalographic (EEG) recordings. 3) The effects of sleep deprivation on the fMRI derived glymphatic flow signal. 4) The effects of the adrenergic antagonist carvedilol on fMRI measurements and sleep intensity. 5) Quantification of cognitive performance before and after a nap in the MRI. Cognitive testing includes: assessments of visual attention, reaction time, paired-associative memory, working memory, emotional recognition and subjective ratings of sleepiness and mood.

DETAILED DESCRIPTION:
Aims and background:

Sleep is a universal biological process. Lack of, or insufficient sleep, has been associated with a range of diseases including obesity, cardiovascular disease, reduced cognition, impaired learning, and increased risk of motor vehicle accidents. Sleep is also associated with neuromolecular alterations in the brain, including reduced firing of arousal maintaining epinephrine and norepinephrine neurons.

A novel molecular function of sleep known as the glymphatic system has recently been described in rodents. This system is specifically activated during non-rapid eye movement (NREM) sleep, and glymphatic flow appear strongly enhanced during sleep when compared to wakefulness. Moreover, it has been shown that adrenergic antagonists enhance glymphatic clearance and flow in rodents. This study aims at applying newly developed functional magnetic resonance imaging (fMRI) protocols to investigate the extent of the glymphatic system non-invasively in humans.

In order for us to quantify the change in glymphatic clearance between sleep and wakefulness, it is necessary to measure the glymphatic process in both vigilance states, requiring that volunteers nap in the MRI scanner. Moreover, to clarify causal relationships, this study will challenge the glymphatic system via adrenergic inhibition. To do so, the investigators will administer the adrenergic antagonist Carvedilol, which can cross the blood-brain barrier. The drug will be perorally administered before a nap in the MRI, in a double blind, placebo controlled manner. To assess sleep quality and function, cognitive testing will be performed before and after the nap in the MRI scanner. Moreover, to distinguish sleep and wakefulness, electroencephalographic (EEG) recordings will be performed during magnetic resonance (MR)-imaging. Because sleep is a strong homeostatic regulated process, sleep quality, duration and timing will be controlled by EEG monitoring, immediately prior to and during the study to ensure that data is intra- and inter-individually comparable.

Hypotheses:

Investigators hypothesis that the fMRI data collected awake and during a nap will be altered by the adrenergic treatment. Specifically, investigator propose the following hypotheses: 1. Sleep promotes cerebrospinal fluid pulsations (glymphatic flow) in the human brain, as measured with fMRI. 2. Challenging the sleep-homeostat by sleep deprivation promotes the fMRI glymphatic flow signal further. 3. The rate of glymphatic flow is expected to be proportional to simultaneously measured non-rapid eye movement EEG slow wave activity. 4: The adrenergic antagonist carvedilol will enhance glymphatic clearance and sleep intensity. 5. The fMRI determined glymphatic flow is associated with improved cognitive performance following sleep. 6. Enhanced glymphatic flow is correlated with enhanced cognitive performance, including: assessments of visual attention, reaction time, paired-associative memory, working memory, emotional recognition and subjective ratings of sleepiness and mood.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer (male or female) between 18 and 35 years.
* Good sleeper with sleep efficiency above 80%.

Exclusion Criteria:

* Current or former primary psychiatric disorder in volunteer of first degree relatives (DSM IV Axis I or WHO ICD-10 diagnostic classification).
* Current or previous neurological disease, severe somatic disease, or the consumption of drugs likely to influence the test results.
* Claustrophobia or fear of being in an MR-scanner.
* Alcohol or drug abuse.
* Regular smoking or nicotine addiction
* Extreme morning or evening type, or extreme short or long sleeper.
* Disordered sleep, regular shift-work or extreme tiredness (e.g. Epworth Sleepiness Scale (ESS) > 10).
* Crossing of multiple time zones within the last 6 months.
* Extreme use of stimulants such as caffeine.
* Not adhering to the prescribed sleep-wake schedule before study initiation.
* Left handedness.
* Obesity (BMI > 27.5).
* Non-fluent in Danish or pronounced visual or auditory impairments.
* Current or past learning disability.
* Large head size (>59 cm in circumference).
* Pregnancy
* Contraindications for MRI (pacemaker, metal implants, etc.).
* Allergy to the ingredients in the administered drug.
* Abnormal ECG (e.g. prolonged QT syndrome, etc.)
* Dizzy when changing from supine to upright position (e.g. postural orthostatic tachycardia syndrome).
* Mild hypotension (blood pressure below 100/70 mmHg)
* Hypertension (blood pressure above 140/90 mmHg).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Measure the change in functional Magnetic Resonance Imaging (fMRI)-detected glymphatic flow in wakefulness and sleep at baseline | Baseline compared to baseline - within same 1 day
Measure and compare functional Magnetic Resonance Imaging (fMRI)-detected glymphatic flow in baseline sleep and in sleep-deprived sleep | Baseline to follow-up 5±3 days
Measure and compare fMRI-detected glymphatic flow in placebo and carvedilol condition | Placebo compared to treatment 5±3 days apart.
Correlate fMRI-detected glymphatic flow with simultaneous detected EEG sleep slow wave activity | Nocturnal sleep compared to sleep during Magnetic Resonance scans within same 1 day.
Measure EEG slow wave activity during Magnetic Resonance imaging and compare Carvedilol with placebo to see how sleep is affected by the treatment | Placebo compared to treatment 5±3 days apart.
Measure if fMRI-detected glymphatic flow correlates with subjective sleepiness ratings | Measurements collected within the same 1 day
Measure fMRI-detected glymphatic flow and whether it correlates with cognitive performance before and after MR imaging | Measurements collected within the same 1 day
Measure fMRI-detected glymphatic flow and whether correlates with changes in cognitive performance from before to after MR imaging | Measurements collected within the same 1 day
Measure whether Carvedilol improves sleepiness after the MR scan compared to placebo | Measurements collected within the same 1 day
Measure whether Carvedilol improves cognitive performance (measurement: psychomotor vigilance test) after the MR scan compared to placebo | Measurements collected within the same 1 day

SECONDARY OUTCOMES:
Measure whether fMRI-detected glymphatic flow is spatially correlated with simultaneous EEG NREM slow wave activity | Measurements collected within the same 1 day
Measure whether fMRI-detected glymphatic flow correlates with simultaneous NREM EEG activity | Measurements collected within the same 1 day
Measure whether fMRI-detected glymphatic flow is positively correlated with sleep driven structural changes in T2 and diffusion weighted (DWI) images | Measurements collected within the same 1 day
Measure whether Carvedilol modulates nocturnal recovery sleep (measurement: EEG slow wave activity) after sleep deprivation | Baseline to follow-up 5±3 days
Measure whether the psychomotor vigilance test is modulated by carvedilol | Placebo compared to treatment 5±3 days apart.
Measure whether the visual attention (measurement: Theory of Visual Attention task) is modulated by carvedilol | Placebo compared to treatment 5±3 days apart.
Measure whether the visual attention (measurement: Theory of Visual Attention task) is modulated by sleep-deprivation | Baseline to follow-up 5±3 days
Measure whether emotional memory performance (measurement: emotional word pair task) is modulated by carvedilol | Placebo compared to treatment 5±3 days apart.
Measure whether emotional memory performance (measurement: emotional word pair task) is modulated by sleep-deprivation | Baseline to follow-up 5±3 days

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian C Sebastian, PhD, Principal Investigator — Neurobiology Research Unit, Rigshospitalet
Locations (1):
- Neurobiology Research Unit, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Via database of Center for Integrated Molecular Brain Imaging (Knudsen et al 2016, NeuroImage). Data will be available for neuroscience research community contingent on approval by scientific board.
Supporting Information: Study Protocol
Time Frame: Data will be made available upon data-analyses completion, about year: 2020.
Access Criteria: Data can be accessed via website or by contacting the NRU lab. Mainly research teams in Europe are granted access.
URL: http://cimbi.dk/